CLINICAL TRIAL: NCT01145547
Title: The Effect of Glycemic Index on Post-prandial Glycemia (Breakfast vs. Lunch) in Patients With Type 1 Diabetes: Quantification With Continuous Glucose Monitoring
Brief Title: Continuous Glucose Monitoring to Measure Effect of Glycemic Index
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Legacy Health System (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Principal Investigator, W. Kenneth Ward, Senior Scientist, Legacy Health System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: kw01
Record Dates: First submitted 2010-06-15; First posted 2010-06-16 (Estimated); Results first posted 2015-10-05 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: glycemic index; Diabetes Mellitus; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low glycemic index effect on post-prandial peak (Active Comparator): Seven adult subjects with type 1 diabetes participated in two experiments, each consisting of two meals each. In one experiment, both meals had a low Glycemic Index.
  Interventions: Device: Dexcom Seven® Plus Continuous Glucose Monitoring sensor
- high glycemic index effect on post-prandial peak (Active Comparator): Seven adult subjects with type 1 diabetes participated in two experiments, each consisting of two meals each. In one experiment, both meals had a high Glycemic Index.
  Interventions: Device: Dexcom Seven® Plus Continuous Glucose Monitoring sensor

INTERVENTIONS:
Device: Dexcom Seven® Plus Continuous Glucose Monitoring sensor — A Dexcom Seven® Plus Continuous Glucose Monitoring sensor was inserted subcutaneously into each subject.

SUMMARY:
Background: Post-prandial hyperglycemia is common in people with type 1 diabetes.

Objective: The aim was to determine the impact of low vs high glycemic index (GI) on post-prandial glycemia for breakfast vs lunch and to quantify these effects with continuous glucose monitoring.

Design: Seven adult subjects with type 1 diabetes participated in two experiments, each consisting of two meals each. In one experiment, both meals had a low GI; in the other, high GI. Meals were given 195 minutes apart and were matched for carbohydrate, protein, and fat content. Each subject received his usual pre-prandial insulin dosage, followed by a continuous subcutaneous basal insulin infusion for the remainder of the experiment. Arterialized venous glucose was analyzed every 15 minutes and sensor glucose was recorded every 5 minutes.

DETAILED DESCRIPTION:
A total of 14 diet studies (each with two meals) were completed in three men and four women. All subjects completed two diet studies in which two meals were served 195 minutes apart. On one study day, two high GI (> 75) meals were given, and on the other study day, two low GI (< 30) meals were given. The low GI and high GI meals were matched for amount of carbohydrates, protein, and fat based on a weight-maintaining diet for each subject. The order of the study treatment (high or low GI) was randomized. Subjects were not informed as the GI of any meal.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of type 1 diabetes mellitus
* patients on insulin pump therapy

Exclusion Criteria:Any patient who was

* pregnancy
* cardiovascular, cerebrovascular, kidney, or liver disease
* uncontrolled chronic medical conditions
* oral or parenteral corticosteroid use
* immunosuppressant use
* visual or physical impairments that impede the use of a continuous glucose monitoring device
* insulin or glucagon allergy
* hypoglycemia unawareness
* requirement of greater than 200 units of insulin per day
* gastroparesis
* any prior gastric surgery
* an allergy to any food items served.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-04; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: W K Ward, MD, Principal Investigator — Legacy Health System
Locations (1):
- Legacy Health System--Holladay Park Campus, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seven subjects with Type 1 diabetes mellitus on subcutaneous insulin pump therapy were recruited from clinics in Portland, Oregon, USA.
Groups:
- Low Glycemic Index, High Glycemic Index: Seven adult subjects with type 1 diabetes participated in two experiments, each consisting of two meals each. In this arm, subjects completed the first study consuming meals with low glycemic index followed by a second study consuming meals with a high glycemic index
  Dexcom Seven® Plus Continuous Glucose Monitoring sensor: A Dexcom Seven® Plus Continuous Glucose Monitoring sensor was inserted subcutaneously into each subject.
- High Glycemic Index, Low Glycemic Index: Seven adult subjects with type 1 diabetes participated in two experiments, each consisting of two meals each. In this arm, subjects completed the first study consuming meals with high glycemic index followed by a second study consuming meals with a low glycemic index
  Dexcom Seven® Plus Continuous Glucose Monitoring sensor: A Dexcom Seven® Plus Continuous Glucose Monitoring sensor was inserted subcutaneously into each subject.
Period: Overall Study
Arm/Group | Low Glycemic Index, High Glycemic Index | High Glycemic Index, Low Glycemic Index
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Seven adult subjects with type 1 diabetes participated in two experiments, each consisting of two meals each. In one experiment, both meals had a low Glycemic Index and in one experiment, both meals had a high Glycemic Index.
  Dexcom Seven® Plus Continuous Glucose Monitoring sensor: A Dexcom Seven® Plus Continuous Glucose Monitoring sensor was inserted subcutaneously into each subject.
Arm/Group | All Study Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Area Under the Curve for Rise in Breakfast Post-prandial.
Description: Arterialized blood glucose was monitored at 15 minute intervals and sensed glucose was recorded at five minute intervals. Mean area under the curve was calculated over the 3 hour period after breakfast for both the high and low glycemic breakfast meals.
Time Frame: Mean area under the curve was calculated at 0, 15min, 30 min, 45 min, 60min, 75 min, 90 min, 105 min, 120min, 135min, 150min, 165min and 180 min after breakfast
Measure: Mean (Standard Deviation); unit: min x (mmol/l)
Arm/Group | Low Glycemic Index Effect on Post-prandial Peak | High Glycemic Index Effect on Post-prandial Peak
Number analyzed (Participants) | 7 | 7
min x (mmol/l) | 61 (135) | 583 (113)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Low Glycemic Index Effect on Post-prandial Peak | High Glycemic Index Effect on Post-prandial Peak
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes